CLINICAL TRIAL: NCT04126928
Title: Validation of PUFA Index in Assessing Untreated Dental Caries Among Malaysian Adult Subpopulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Amy Liew, Lecturer, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UKM 1.5.3.5/244/DD/2015/008(2)
Record Dates: First submitted 2019-10-09; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Pulpitis; Apical Periodontitis
Keywords: orthopantomograph; periapical index; reliability; sensitivity; specificity
MeSH Terms: conditions — Pulpitis; Periapical Periodontitis; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant (Other): Each participant will go through (i) screening using DMFT and PUFA, (ii) orthopantomography assessment using PAI, and (iii) comprehensive clinical examination to derive pulpal and periapical diagnoses
  Interventions: Diagnostic Test: Screening using DMFT and PUFA, orthopantomogram is taken and assessed using PAI, comprehensive clinical examination to diagnose pulpal and periapical conditions.

INTERVENTIONS:
Diagnostic Test: Screening using DMFT and PUFA, orthopantomogram is taken and assessed using PAI, comprehensive clinical examination to diagnose pulpal and periapical conditions.

SUMMARY:
PUFA Index was introduced to detect the clinical consequences of untreated dental caries. To date, there are no studies on the reliability and accuracy of the PUFA index as a screening tool. Other than indices, radiographs were sometimes used as a screening tool using the validated Periapical Index (PAI). The aim of this study was to evaluate the reliability and accuracy of PUFA and PAI in screening for clinical outcomes of untreated caries, specifically pulpal and periapical diseases. The reference standard is the clinical diagnosis, as categorized by the American Association of Endodontists. Intra- and inter-examiner reliability will be determined using Cohen's kappa. Sensitivity, specificity, positive predictive value, and negative predictive value will be calculated. Receiver Operating Characteristics (ROC) contrast estimation will be computed to compare the two index tests.

DETAILED DESCRIPTION:
The index of decayed-missing-filled permanent teeth (DMFT) records decayed (D), missing (M), or filled (F) teeth in an individual, but it fails to give information about the clinical outcomes of untreated dental caries. A new index complements the DMFT index by recording the advancement of the caries lesion into surrounding tissues, including pulpal involvement (P), ulceration due to tooth fragments (U), fistula formation (F) and abscess (A). The PUFA index has yet to be validated in the adult population. Other than indices, radiographs were sometimes used as a screening tool using the validated Periapical Index (PAI). Hence, the aim of this study is to evaluate the reliability and accuracy of PUFA and PAI in screening for clinical outcomes of untreated caries, specifically pulpal and periapical diseases. The study will be carried out in Primary Care Clinic, Faculty of Dentistry, Universiti Kebangsaan Malaysia. Consecutive sampling will be used; all eligible patients are invited to participate. The inclusion criteria are as follow:

i. New patient, not receiving active dental treatment at the time of study ii. Adult patient (18 years old or above) iii. Having at least 12 teeth in the oral cavity iv. Presented with the clinical situation for which radiograph(s) were indicated v. No radiograph was taken within the last six months The reference standard is the clinical diagnosis, as categorized by the American Association of Endodontists. A comprehensive examination will be carried out for each tooth, followed by investigation using orthopantomography (OPG), periapical radiograph, periodontal probing, heat test, cold test, electric pulp tester when indicated, to aid in arriving at the definitive diagnosis.

Two independent, trained dentists are employed to screen the participants using DMFT and PUFA indices, blinded to the clinical diagnosis and PAI scoring. The examination is done using only a mouth mirror.

Another two independent, trained dentists, blinded to the clinical diagnoses and the PUFA scoring, will score each tooth on the orthopantomograph for the periapical status using the Periapical Index (PAI).

The outcome of PUFA is dichotomized as Positive (PUFA>0) or Negative (PUFA=0) for each tooth. Similarly, the PAI was dichotomized as Positive (PAI≥3) or Negative (PAI<3). Intra- and inter-examiner reliability will be determined using Cohen's kappa. Sensitivity, specificity, positive predictive value, and negative predictive value will be calculated. ROC contrast estimation will be computed to compare the two index tests.

ELIGIBILITY:
Inclusion Criteria:

* New patient, not receiving active dental treatment at the time of the study
* Adult patient (18 years old or above)
* Has at least 12 teeth in the oral cavity
* Presented with the clinical situation for which radiograph(s) were indicated (American Dental Association 2012)
* No radiograph was taken within the last 6 months

Exclusion Criteria:

* Pregnant
* Medically compromised (American Society of Anesthesiologists ASA3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
DMFT | All variables for each person are collected at one point in time. An average visit is two hours per person.
  Decayed (D), missing (M), or filled (F) tooth, assessed clinically using only mouth mirror
PUFA | All variables for each person are collected at one point in time. An average visit is two hours per person.
  Pulpal involvement (P), ulceration due to tooth fragments (U), fistula formation (F) and abscess (A), assessed clinically using only mouth mirror
Periapical Index (PAI) | All variables for each person are collected at one point in time. An average visit is two hours per person.
  An ordinal scale of 5 scores ranging from 1 (healthy) to 5 (severe apical periodontitis), assessed radiographically. Higher scores mean a worse outcome.
Diagnosis of pulpal and periapical diseases | All variables for each person are collected at one point in time. An average visit is two hours per person.
  Diagnosis of pulpal and periapical diseases using the diagnostic criteria of American Association of Endodontists following comprehensive clinical examination

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Abdullah, MClinDent, Principal Investigator — National University of Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glickman GN. AAE Consensus Conference on Diagnostic Terminology: background and perspectives. J Endod. 2009 Dec;35(12):1619-20. doi: 10.1016/j.joen.2009.09.029. No abstract available. PMID 19932336
- [Background] Monse B, Heinrich-Weltzien R, Benzian H, Holmgren C, van Palenstein Helderman W. PUFA--an index of clinical consequences of untreated dental caries. Community Dent Oral Epidemiol. 2010 Feb;38(1):77-82. doi: 10.1111/j.1600-0528.2009.00514.x. Epub 2009 Dec 7. PMID 20002630
- [Background] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698

DOCUMENTS (1):
  • Study Protocol (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT04126928/Prot_000.pdf